CLINICAL TRIAL: NCT01144845
Title: Study of Persistent Postsurgical Pain Following Thoracic Surgery in Patients With Pulmonary Malignancies
Brief Title: Chronic Pain Following Thoracic Surgery
Acronym: PTPS-18
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kasper Grosen, PhD fellow, Master of Health Sciences, RN, University of Aarhus
Other Study IDs: PTPS-18
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pain, Postoperative
Keywords: Thoracotomy; Thoracic Surgery; Thoracic Surgical Procedures; Thoracic Surgery, Video-Assisted; Lung Neoplasms; Thoracic Nerves
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms | interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracic surgical patients: Patients with pulmonary malignancies
  Interventions: Procedure: Thoracic surgery

INTERVENTIONS:
Procedure: Thoracic surgery — Thoracoscopy or anterior thoracotomy

SUMMARY:
Pain that persists after the healing of a surgical wound has previously been described as an important, but often unrecognized clinical problem. Persistent postsurgical (chronic postoperative pain) is the consequence of either ongoing inflammation or more common neuropathic pain as a result of surgical damage to peripheral nerves.

Previous studies have shown that chronic pain is a frequent and serious complication following thoracic surgery. However, the prevalence of chronic pain following both thoracoscopy and anterior thoracotomy in patients with pulmonary malignancies is poorly characterized and the impact of this pain on patients' lives remains unclear. Thus, this study aims to investigate the prevalence of chronic pain following thoracoscopy or anterior thoracotomy, and the severity and impact of persistent post-surgical pain on daily life.

This study is working with several hypotheses: 1.) persistent postsurgical pain following lung cancer surgery is predominantly of neuropathic nature and the presence of neuropathic symptoms increases the severity of postsurgical pain and reduces the patient's quality of life, 2.) the prevalence of chronic pain is reduced over time, and 3.) less invasive thoracic surgical interventions reduces the risk of the development of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who previously underwent thoracic surgery with lung resection from January 2000 to december 2009

Exclusion Criteria:

* Death

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent thoracic surgery due to pulmonary malignancies at the Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Denmark
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Presence of persistent postsurgical pain | Within 10 years after thoracic surgery

SECONDARY OUTCOMES:
Location of persistent postsurgical pain | Within 10 years after thoracic surgery
Duration of postsurgical pain | Within 10 years after thoracic surgery
Course of persistent postsurgical pain | Within 10 years after thoracic surgery
Severity of postsurgical pain | Within 10 years after thoracic surgery
Characteristics of persistent postsurgical pain | Within 10 years after thoracic surgery
Symptoms associated with persistent postsurgical pain | Within 10 years after thoracic surgery
Treatment of and effect of treatment on persistent postsurgical pain | Within 10 years after thoracic surgery
Effect of postsurgical pain on activity, mood, walking ability, work, interpersonal relations, sleep and quality of life | Within 10 years after thoracic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Grosen, PhDS, MHScS, RN, Principal Investigator — Department of Cardiothoracic and Vascular surgery, Aarhus University Hospital, Skejby, Denmark; Hans K Pilegaard, MD, Study Director — Department of Cardiothoracic and Vascular surgery, Aarhus University Hospital, Skejby, Denmark; Vibeke Hjortdal, MD, Professor, DMSc, PhD, Study Chair — Department of Cardiothoracic and Vascular surgery, Aarhus University Hospital, Skejby, Denmark; Mogens P Jensen, MD, PhD, Study Chair — Department of Rheumatology, Aarhus University Hospital, Aarhus Hospital, Denmark
Locations (1):
- Department of Cardiothoracic and Vascular surgery, Aarhus University Hospital, Skejby, Aarhus N, Denmark